CLINICAL TRIAL: NCT02147873
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of Azacitidine With or Without Birinapant With a Single Arm Open-Label Run-In Phase in Subjects With Higher Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Brief Title: Study of Azacitidine With or Without Birinapant in Subjects With MDS or CMMoL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of efficacy
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TL32711-RAN-0094-PTL; 2014-001719-37 (EudraCT Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-28 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML)
Keywords: MDS; CMML; myelodysplastic syndrome; chronic myelomonocytic leukemia; TL32711; TL32711-0094; azacitidine; birinapant; higher risk; naive; double blind; placebo; placebo controlled; randomized
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — birinapant; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azacitidine with birinapant (Active Comparator): Azacitidine 75 mg/m2 IV on days 1-5, 8 & 9 OR days 1-7 and birinapant 13 mg/m2 IV twice a week (days 1 & 4) for 3 out of 4 weeks
  Interventions: Drug: birinapant; Drug: Azacitidine
- Azacitidine and placebo (Placebo Comparator): Azacitidine 75mg/m2 IV days 1-5, 8 & 9 OR days 1-7 and placebo IV twice a week (days 1 & 4) for 3 out of 4 weeks
  Interventions: Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: birinapant
  Other Names: TL32711
  Arms: azacitidine with birinapant
Drug: Azacitidine
Drug: Placebo
  Arms: Azacitidine and placebo

SUMMARY:
This is a randomized double blind placebo controlled study of azacitidine with or without birinapant in subjects with higher risk Myelodysplastic syndrome, secondary MDS or myelomonocytic leukemia (CMMoL) who are naïve, to azacitidine therapy. Pre-clinical and mechanistic studies support that azacitidine may modulate pathways that enable birinapant-mediated anti-tumor activity.

DETAILED DESCRIPTION:
This is a randomized double blind placebo controlled study of azacitidine with or without birinapant in subjects with higher risk Myelodysplastic syndrome, secondary MDS or myelomonocytic leukemia (CMMoL)

The primary purpose of this study is :

-To compare the relative effect of azacitidine plus birinapant versus azacitidine plus placebo on response rate in patients with higher-risk MDS, secondary MDS or CMMoL.

The secondary purpose of this study is to compare effect of azacitidine plus birinapant relative to azacitidine with placebo on:

* Hematologic improvement
* Relapse free survival
* Time to respond
* Change in transfusion requirements
* Duration of response
* Overall survival
* Adverse events

The exploratory objective of this study is to assess exploratory translational biomarkers for antitumor effects.

ELIGIBILITY:
key Inclusion Criteria:

* Morphologically confirmed diagnosis of MDS/CMMoL according to FAB or WHO classification, including RAEB-t and MDS/MPN
* International prognostic score-revised (IPSS-R) of >3.5 (Intermediate, High or Very High)
* Previously untreated with hypomethylating agents for MDS/CMMoL
* Performance status of 0, 1 or 2 by the ECOG scale
* Adequate renal and liver function
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening within 96 hours prior to the first study dose.
* Female subjects of childbearing potential and male subjects with partners of childbearing potential should ensure use of a highly effective method of birth control as defined by the investigator, for example, those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly during the study and for a period of 3 months following the last dose of any drug administered during the study.

Key Exclusion Criteria:

* Relapsed or refractory to hypomethylating agents
* Acute myeloid leukemia (AML), except those patients with RAEB-t who are not candidates for intensive AML therapy.
* Participated in any interventional study within 4 weeks of randomization or 5 half lives (whichever is longer).
* Received any hematopoietic growth factors within 14 days prior to screening.
* Prior malignancy or secondary malignancy within the prior 2 years (except in situ cervical cancer, squamous cell carcinoma or basal cell carcinoma of the skin).
* known diagnosis of human immunodeficiency virus or chronic active Hep B or C.
* Uncontrolled hypertension
* Impaired cardiac function, uncontrolled cardiac arrhythmias despite medications, or clinically significant cardiac disease
* Lack of recovery of prior adverse events to Grade ≤1 severity (National Cancer Institute Common Terminology Criteria for Adverse Events version 4) (except alopecia) due to therapy administered prior to the initiation of study drug dosing.
* Nursing or pregnant.
* Known allergy or hypersensitivity to any of the formulation components
* Any concurrent disease and/or medical condition that, in the opinion of the Investigator, would prevent the subject's participation.
* History of cranial nerve palsy.
* Being treated with anti-TNF therapies or has been treated with an anti-TNF therapy within 5 half-lives of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Response Rate | participants will be followed for until disease progression an expected average of 1 year

SECONDARY OUTCOMES:
Hematologic improvement | participants will be followed for until disease progression an expected average of 1 year
Relapse free survival | An expected average of 2 year post last study dose
  According to modified IWG 2006 criteria
Time to respond | participants will be followed for until disease progression an expected average of 1 year
Change in transfusion requirements | participants will be followed for until disease progression an expected average of 1 year
duration of response | participants will be followed for until disease progression an expected average of 1 year
  According to modified IWG 2006 criteria
overall survival | An expected average of 2 year post last study dose
Adverse events profile | participants will be monitored for adverse events throughout the treatment period and during follow up period

OTHER OUTCOMES:
exploratory translational biomarkers for antitumor effect | 30 days

CONTACTS AND LOCATIONS:
Locations (76):
- United States (46):
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - North County Oncology, Oceanside, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Stanford Hospital and Clinics, Stanford, California
  - Wellness Oncology & Hematology, West Hills, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Bond Clinic PA, Winter Haven, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Simmons Cancer Institute at Southern Illinois University, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville Hospital/James Graham Brown Cancer Center, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Monter Cancer Center, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Carolina Blood and Cancer Care Associates, P.A., Rock Hill, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Tyler Hematology Oncology PA, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Metro South Health, Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - The Alfred, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Perth Blood Institute, Nedlands, Western Australia
- Germany (9):
  - Klinikum der Ludwig-Maximilians-Universitat Munchen, Munich, Bavaria
  - Klinikum Rechts der Isar, Technischen Universitat Munchen, München, Bavaria
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Marien Hospital Dusseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Halle, Halle, Saxony-Anhalt
  - Universitatsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitatsklinik Heidelberg, Heidelberg
  - Universitatsklinikum Wurzburg, Würzburg
- Spain (11):
  - Hospital Germans Trias I Pujol, Badalona, Badalona
  - Hospital University Reina Sofia, Córdoba, Cordoba
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Gregorio Maranon, Madrid, Madrid
  - MD Anderson Cancer Center, Madrid, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, S/C Tenerife
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Complejo Hospitalario Virgen de la Salud, Toledo, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia